CLINICAL TRIAL: NCT03469271
Title: Resistance Training and 1,25 (OH)2D3 Administration to Maintain Respiratory Muscle Function and Reduce Pneumonia Risk in Cancer Patients
Brief Title: Maintain Respiratory Muscle Function and Reduce Pneumonia Risk in Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Andersen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 17-009440
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Pneumonia
MeSH Terms: conditions — Neoplasms; Pneumonia | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Training and Placebo (Other): Inspiratory isometric resistance training with the Threshold Inspiratory Muscle Trainer (IMT) plus oral placebo for eight weeks
  Interventions: Other: Inspiratory isometric resistance training; Drug: Oral Placebo; Device: Threshold Inspiratory Muscle Trainer (IMT)
- Sham Training and Vitamin D3 Metabolite (Other): Sham inspiratory isometric resistance training with the Threshold Inspiratory Muscle Trainer (IMT) plus 1,25 (OH)2 D3 orally for eight weeks
  Interventions: Drug: 1,25 (OH)2 D3; Other: Sham Inspiratory Isometric Resistance Training; Device: Threshold Inspiratory Muscle Trainer (IMT)
- Training and Vitamin D3 Metabolite (Other): Inspiratory isometric resistance training with the Threshold Inspiratory Muscle Trainer (IMT) plus 1,25(OH)2 D3 orally for eight weeks
  Interventions: Drug: 1,25 (OH)2 D3; Other: Inspiratory isometric resistance training; Device: Threshold Inspiratory Muscle Trainer (IMT)
- Sham Training and Placebo (Other): Sham inspiratory isometric resistance training with the Threshold Inspiratory Muscle Trainer (IMT) plus oral placebo orally for eight weeks
  Interventions: Drug: Oral Placebo; Other: Sham Inspiratory Isometric Resistance Training; Device: Threshold Inspiratory Muscle Trainer (IMT)

INTERVENTIONS:
Drug: 1,25 (OH)2 D3 — 0.25 micrograms, taken daily for eight weeks, orally
  Other Names: Calcitriol; 1, 25-dihydroxycholecalciferol; Rocaltrol
  Arms: Sham Training and Vitamin D3 Metabolite; Training and Vitamin D3 Metabolite
Other: Inspiratory isometric resistance training — A small hand-held reusable device to increase muscle strength and endurance through inhalation therapy. Participants will inhale through a valve which provides resistance that increases the work of breathing and exercises the respiratory muscles.Participants in the active groups will breathe against a resistance set to generate 30% of maximal inspiratory pressure (PImax).
  Arms: Training and Placebo; Training and Vitamin D3 Metabolite
Drug: Oral Placebo — Placebo will be created to mimic the appearance of the study drug
  Arms: Sham Training and Placebo; Training and Placebo
Other: Sham Inspiratory Isometric Resistance Training — A small hand-held reusable device to increase muscle strength and endurance through inhalation therapy. Participants will inhale through a valve which provides resistance that increases the work of breathing and exercises the respiratory muscles. Participants in the sham group will train daily against a resistance set to only 15% PImax.
  Arms: Sham Training and Placebo; Sham Training and Vitamin D3 Metabolite
Device: Threshold Inspiratory Muscle Trainer (IMT) — A small hand-held reusable device to increase muscle strength and endurance through inhalation therapy. Participants will inhale through a valve which provides resistance that increases the work of breathing and exercises the respiratory muscles.
  Other Names: Threshold IMT Breathing Trainer

SUMMARY:
This research is intended to begin to explore the impact of inspiratory muscle resistance exercise and/or 1,25(OH)2D3 for improving respiratory muscle strength in cancer patients (subjects).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Renal and hepatic function (creatinine </= 2 x the institutional upper limit of normal; bilirubin </= 2 x the institutional upper limit of normal)
* No contraindication to receive either of the planned interventions of inspiratory resistance training or 1,25(OH)2D3 in the opinion of the healthcare provider
* No difficulties with swallowing oral medications in the opinion of the enrolling physician

Exclusion Criteria:

* Patient is taking calcium or Vitamin D supplements and is unwilling to stop for 8 weeks
* Severe chronic obstructive pulmonary disease (oxygen dependent or patient self-reports unable to walk one block without difficulty)
* Calcium or phosphorus level above the institutional upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A study coordinator worked closely with Dr. Jatoi in numerous clinics in the Division of Medical Oncology to identify potential candidates for this study.
Pre-assignment Details: Nothing to report
Period: Overall Study
Arm/Group | Training and Placebo | Sham Training and Vitamin D3 Metabolite | Training and Vitamin D3 Metabolite | Sham Training and Placebo
Started | 16 | 15 | 15 | 17
Completed | 14 | 15 | 15 | 16
Not Completed | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Training and Placebo | Sham Training and Vitamin D3 Metabolite | Training and Vitamin D3 Metabolite | Sham Training and Placebo | Total
Number analyzed (Participants) | 16 | 15 | 15 | 17 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 11 | 15 | 51
  >=65 years | 3 | 3 | 4 | 2 | 12
Age, Continuous [Mean (Full Range); unit: years] | 52.5 [34 to 72] | 58 [42 to 81] | 55 [31 to 74] | 51 [26 to 75] | 54 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 13 | 12 | 50
  Male | 3 | 3 | 2 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 15 | 16 | 60

OUTCOME MEASURES:

1. Primary Outcome: Sniff Nasal Inspiratory Pressure (SNIP)
Description: SNIP is a test of maximal inspiratory muscle force exerting from the diaphram. Patients sniff forcefully through one nostril while the other is obstructed. The best of 10 measurements is recorded.
Time Frame: 8 weeks
Population: Patients completing all 8 weeks of treatment.
Measure: Mean (Full Range); unit: cmH20
Arm/Group | Training and Placebo | Sham Training and Vitamin D3 Metabolite | Training and Vitamin D3 Metabolite | Sham Training and Placebo
Number analyzed (Participants) | 14 | 15 | 15 | 16
cmH20 | 90 [51 to 190] | 87 [51 to 159] | 89 [43 to 150] | 109 [74 to 153]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Training and Placebo | Sham Training and Vitamin D3 Metabolite | Training and Vitamin D3 Metabolite | Sham Training and Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03469271/Prot_SAP_000.pdf